CLINICAL TRIAL: NCT02875262
Title: Deferoxamine in Aneurysmal Subarachnoid Hemorrhage Trial
Acronym: DASH
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Radboud University Medical Center (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL58448.091.16
Record Dates: First submitted 2016-07-20; First posted 2016-08-23 (Estimated); Last update posted 2023-04-24 (Actual); Status verified 2023-04

CONDITIONS: Intracranial Aneurysm; Subarachnoid Hemorrhage
Keywords: intracranial aneurysm; subarachnoid hemorrhage; stroke; chelator
MeSH Terms: conditions — Intracranial Aneurysm; Subarachnoid Hemorrhage; Stroke | interventions — Deferoxamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients will be given deferoxamine 32 mg/kg/day (max iv rate 15 mg/kg/hr), patients with ferritin levels between 2,000 and 3,000 ng/ml will receive 32 mg/kg/day and patients with serum ferritin levels below 2,000 ng/ml wil receive 25 mg/kg/day. duration 3 days
  Interventions: Drug: Deferoxamine
- placebo (Placebo Comparator): NaCl 0.9% in similar dosis to treatment arm
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Deferoxamine — Patients will be given deferoxamine 32 mg/kg/day (max iv rate 15 mg/kg/hr), patients with ferritin levels between 2,000 and 3,000 ng/ml will receive 32 mg/kg/day and patients with serum ferritin levels below 2,000 ng/ml wil receive 25 mg/kg/day.during 3 days
  Other Names: desferal
  Arms: Treatment
Other: placebo — placebo (NaCl 0.9%) in equal dose to treatment
  Arms: placebo

SUMMARY:
Aneurysmal subarachnoid hemorrhage (SAH) is a form of stroke in which secondary neurological deterioration is an important cause of mortality and morbidity. These secondary changes, so called delayed cerebral ischemia (DCI), are caused by lysis of erythrocytes which can react to form iron, an toxic substance to the brain. Iron chelators remove the excess of iron and are standard care in iron-overloaded patients. Deferoxamine (DFO) an chelator has not been evaluated in SAH patients. This study evaluates the safety of deferoxamine in SAH patients.

DETAILED DESCRIPTION:
Aneurysmal subarachnoid hemorrhage (SAH) is a devastating form of stroke affecting relatively young patients. It has an incidence of about 7 per 100,000. Associated economic costs are high. Treatment of the aneurysm to prevent rebleeding is the primary goal. Nevertheless, 3 to 12 days after the initial bleeding secondary ischemic changes occur in 30% of the patients. This delayed cerebral ischemia (DCI) remains the most important cause of mortality and morbidity in patients surviving aneurysm treatment.

Aneurysmal SAH exposes the brain to erythrocytes. Several days after the hemorrhage lysis of erythrocytes takes place and the brain is exposed to high concentrations of hemoglobin. Elevated hemoglobin concentrations are present not only at the basal surface of the brain, but also distributed around the brain and into deeper layers of the cortex. Heme is degraded by heme-oxygenase into carbon monoxide, biliverdin and iron. Free iron can react with H2O and O2- to form hydroxyl radicals (OH*). The generation of hydroxyl radicals in this cascade, known as the Haber-Weiss or Fenton reaction, leads to extraction of hydrogen from unsaturated lipids in the cell membrane and initiates lipid peroxidation. Additionally it can exacerbate excitotoxicity by increased intracellular iron accumulation.

Iron chelators remove the excess of iron and are standard care in iron-overloaded patients. The use of iron chelators for SAH has been subject of animal studies with promising results on reduced vasospasm, oxidative stress, neuronal cell death and mortality. No clinical study for the use of deferoxamine in aneurysmal subarachnoid hemorrhage has been performed. A safety study for the use of Deferoxamine in patients in intracerebral hemorrhage (which is distinct from subarachnoid hemorrhage) has been performed. There were no associated serious adverse events or mortality, Deferoxamine is a chelator is used for more than 40 years in patients with iron overload diseases. This study investigates the safety and tolerability of deferoxamine versus placebo in patients with SAH for 3 consecutive days.

ELIGIBILITY:
Inclusion Criteria:

* subarachnoid hemorrhage diagnosed by CT on admission,
* Randomizable within 72 hours of subarachnoid hemorrhage,
* Saccular intracranial aneurysm proven by cerebral angiography or CTA,
* Surgical or endovascular obliteration is performed,
* Able to obtain written informed consent from patient or surrogate.
* Patients in a good clinical grade (WFNS 1-3)

Exclusion Criteria:

* Pregnancy, as confirmed by routine urine test on admission,
* Abnormal renal function at time of randomization (GFR <60 mL/min)
* Elevated liver function test at time of randomization (AST > 45 U/L and ALT > 35 U/L.)
* History of liver disease or active liver disease, Active renal disease,
* Hypersensitivity to deferoxamine,
* Patient taking medication not recommended for concomitant use with deferoxamine as per the product label (e.g. high dose vit. C medication).
* Patients not able to complete the study follow-up the presence of 4 or more of the following exclusion criteria (risk modifiers for ARDS):

  * Tachypnea (respiratory rate >30)
  * SpO2 <95%
  * Obesity (BMI >30)
  * Acidosis (pH <7.35)
  * Hypoalbuminemia (albumin <3.5 g/dL)
  * concurrent use of chemotherapy

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-12-02 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
safety (drug related adverse events; i.e. renal and hepatic dysfunction) | 6 months
  drug related adverse events; i.e. renal and hepatic dysfunction, ARDS

SECONDARY OUTCOMES:
efficacy (new cerebral ischemia compared between intervenation and placebo) | 6 months
  number of patients with delayed cerebral ischemia, which is defined by new, not treatment related cerebral ischemia as registered on CT or MR imaging

CONTACTS AND LOCATIONS:
Overall Officials: Jeroen Boogaarts, M.D., Ph.D., Principal Investigator — Radboud University Medical Center
Locations (2):
- Netherlands (2):
  - Radboudumc, Nijmegen, Gelderland
  - University Medical Center Groningen, Groningen

IPD SHARING:
Plan to Share IPD: Yes
core data will be published

REFERENCES:
- [Derived] Van der Loo LE, Aquarius R, Teernstra O, Klijn K, Menovsky T, van Dijk JMC, Bartels R, Boogaarts HD. Iron chelators for acute stroke. Cochrane Database Syst Rev. 2020 Nov 24;11(11):CD009280. doi: 10.1002/14651858.CD009280.pub3. PMID 33236783